CLINICAL TRIAL: NCT00049569
Title: Intensive Induction Therapy for Children With Acute Lymphoblastic Leukemia (ALL) Who Experience a Bone Marrow Relapse
Brief Title: Combination Chemotherapy and Imatinib Mesylate in Treating Children With Relapsed Acute Lymphoblastic Leukemia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-01798; NCI-2012-01798 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); COG-AALL01P2; CDR0000258120; AALL01P2 (Other: Children's Oncology Group); AALL01P2 (Other: CTEP); U10CA098543 (NIH)
Record Dates: First submitted 2002-11-12; First posted 2003-01-27 (Estimated); Last update posted 2013-10-08 (Estimated); Status verified 2013-10

CONDITIONS: L1 Childhood Acute Lymphoblastic Leukemia; L2 Childhood Acute Lymphoblastic Leukemia; Non-T, Non-B Childhood Acute Lymphoblastic Leukemia; Recurrent Childhood Acute Lymphoblastic Leukemia; T-cell Childhood Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Cytarabine; Methotrexate; Vincristine; Prednisone; pegaspargase; Doxorubicin; Imatinib Mesylate; Cyclophosphamide; Etoposide; Filgrastim; Leucovorin; Asparaginase; Hydrocortisone

ARMS (2):
- Arm I (Experimental): See detailed description.
  Interventions: Drug: cytarabine; Drug: methotrexate; Drug: vincristine sulfate; Drug: prednisone; Drug: pegaspargase; Drug: doxorubicin hydrochloride; Drug: imatinib mesylate; Drug: cyclophosphamide; Drug: etoposide; Biological: filgrastim; Drug: leucovorin calcium; Drug: asparaginase
- Arm II (Experimental): See detailed description.
  Interventions: Drug: cytarabine; Drug: methotrexate; Drug: vincristine sulfate; Drug: prednisone; Drug: pegaspargase; Drug: doxorubicin hydrochloride; Drug: imatinib mesylate; Drug: cyclophosphamide; Drug: etoposide; Biological: filgrastim; Drug: leucovorin calcium; Drug: asparaginase; Drug: therapeutic hydrocortisone

INTERVENTIONS:
Drug: cytarabine — Given IT
Drug: methotrexate — Given IT
Drug: vincristine sulfate — Given IV
Drug: prednisone — Given PO
Drug: pegaspargase — Given IM
Drug: doxorubicin hydrochloride — Given IV
Drug: imatinib mesylate — Given PO
Drug: cyclophosphamide — Given IV
Drug: etoposide — Given IV
Biological: filgrastim — Given SC
Drug: leucovorin calcium — Given IV
Drug: asparaginase — Given IM
Drug: therapeutic hydrocortisone — Given IT
  Arms: Arm II

SUMMARY:
Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Imatinib mesylate may stop the growth of cancer cells by blocking the enzymes necessary for cancer cell growth. Combining more than one chemotherapy drug with imatinib mesylate may kill more cancer cells. Randomized phase II trial to study the effectiveness of combination chemotherapy and imatinib mesylate in treating children who have relapsed acute lymphoblastic leukemia.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the feasibility and safety of using an intensified sequential induction regimen to treat children with acute lymphoblastic leukemia (ALL), who experience an isolated, or combined bone marrow relapse.

II. To determine the potential of this regimen to serve, as a backbone, for the future testing of novel therapeutic agents.

SECONDARY OBJECTIVES:

I. To estimate the remission re-induction rates and four-month event-free survival (EFS) for children, stratified by the duration of first remission.

II. To determine the feasibility of measuring minimal residual disease (MRD) quantitatively in all patients at time points throughout re-induction, and to correlate post-remission events with disease burden during induction.

III. To use deoxyribonucleic acid (DNA) arrays to characterize patterns of gene expression that predict treatment failure, and to compare gene expression profiles at the time of relapse with those at the time of initial diagnosis to gain an understanding of the pathways that may be involved in disease recurrence.

IV. To determine the feasibility of combining intensive re-induction therapy with imatinib mesylate (STI571) for children with a relapse of Philadelphia chromosome positive (Ph+) ALL.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM I:

Treatment Block 1: Patients receive cytarabine intrathecally (IT) on day 1 and methotrexate IT on days 15 and 29. Patients also receive vincristine intravenously (IV) on days 1, 8, 15, and 22; prednisone orally (PO) twice or thrice daily (BID or TID) on days 1-29; pegaspargase intramuscularly (IM) on days 2, 8, 15, and 22; and doxorubicin IV over 15 minutes on day 1. Ph-positive patients also receive imatinib mesylate PO on days 1-14.

Treatment Block 2: Patients receive methotrexate IT on days 1 and 22, cyclophosphamide IV over 30 minutes and etoposide IV over 2 hours on days 1-5, and filgrastim (G-CSF) subcutaneously (SC) beginning on day 6 and continuing until blood counts recover. Patients also receive methotrexate IV over 24 hours on day 22 followed by leucovorin calcium IV every 6 hours on days 24 and 25. Ph-positive patients receive imatinib mesylate PO on days 1-14.

Treatment Block 3a (Ph-negative patients): Patients receive cytarabine IV over 3 hours every 12 hours on days 1, 2, 8, and 9, asparaginase IM on days 2 and 9, and G-CSF SC beginning on day 10 and continuing until blood counts recover.

Treatment Block 3b (Ph-positive patients): Patients receive cytarabine IV over 3 hours every 12 hours on days 1 and 2, asparaginase IM on day 2, and G-CSF SC beginning on day 3 and continuing until blood counts recover. Patients also receive imatinib mesylate PO on days 1-14.

ARM II:

Treatment Block 1: Patients receive cytarabine IT on day 1 and then methotrexate, cytarabine and hydrocortisone IT (triple intrathecal therapy; TIT) on days 8, 15, 22, and 29. Vincristine, prednisone, pegaspargase, doxorubicin, and imatinib mesylate are administered as in arm I.

Treatment Block 3: Patients receive cytarabine, asparaginase, G-CSF, and imatinib mesylate as in arm I.

Treatment Block 2: Patients receive TIT on days 1 and 22. Patients then receive cyclophosphamide, etoposide, G-CSF, methotrexate IV, leucovorin calcium, and imatinib mesylate as in arm I. After each block is completed, disease is assessed. The next block is started on day 36 if blood counts have recovered and marrow during block 1 is at least M2/M3. Patients are removed from protocol therapy if disease progresses, unacceptable toxicity occurs, marrow is M2/M3 at day 15 of the second administered block of treatment, or cerebrospinal fluid blasts persist after 6 weekly doses of TIT.

After completion of study treatment, patients are followed up for 4 months.

PROJECTED ACCRUAL: A total of 63-126 patients will be accrued for this study within 14 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients with acute lymphoblastic leukemia (ALL) in first relapse involving the bone marrow (M3 marrow), with or without associated extramedullary disease; this includes patients who are Philadelphia chromosome-positive
* Shortening fraction of >= 28% by echocardiogram, or ejection fraction of >= 50% by gated radionuclide study
* Cumulative prior anthracycline exposure of =< 350 mg/m^2 (each 10 mg/m^2 dose of idarubicin should be calculated as the isotoxic equivalent of 50 mg/m^2 of daunorubicin or adriamycin)
* All patients and/or their parents or legal guardians must sign a written informed consent
* All institutional, Food and Drug Administration (FDA), and National Cancer Institute (NCI) requirements for human studies must be met

Exclusion Criteria:

* Patients with B-cell ALL (L3 morphology or evidence of myc translocation by molecular or cytogenetic technique) are not eligible
* Patients with Down syndrome are excluded due to the administration of methotrexate in Block 2
* Patients who have undergone prior stem cell transplantation (SCT) are ineligible if:

  * They received SCT less than 12 months prior to study entry
  * They are still receiving immunosuppression for the treatment of graft-versus-host disease (GVHD)
  * They have active fungal infection at time of study entry
  * They have had invasive filamentous fungal infection at any time post-SCT
* Pregnant or lactating females are ineligible as the medications used in this protocol could be harmful to unborn children and infants
* Patients with prior isolated extramedullary relapse are ineligible

Ages: 1 Year to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 126 (Estimated)
Dates: Start 2003-01; Primary Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
Feasibility assessed by excessive early deaths, induction failures, and early relapses | Up to 4 months
Toxicity assessed using CTC version 2.0 | Up to 4 months
  Will be tabulated in detail.

SECONDARY OUTCOMES:
Overall remission reinduction (CR2) rate | Up to 4 months
EFS | 4 months
  The Kaplan-Meier method will be used.
MRD | Up to 4 months
  The percentage of MRD positive patients will be estimated at the end of each block. Cox regression will be utilized to correlate MRD values with EFS.
Feasibility of combining intensive re-induction therapy with imatinib mesylate | Up to 4 months
  Will be determined using descriptive statistics due to the small sample size.
Percentage of patients who were able to complete the triple re-induction therapy with imatinib mesylate | Up to 4 months
  Will be estimated.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Raetz, Principal Investigator — Children's Oncology Group
Locations (1):
- Children's Oncology Group, Arcadia, California, United States